CLINICAL TRIAL: NCT05896280
Title: Effects of Endoclip Papilloplasty and Relationship Between Post-operative Microecological Environment and Recurrent Bile Duct Stones
Brief Title: Effect of ECPP on Recurrent Bile Duct Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LM2023425
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-10

CONDITIONS: Sphincterotomy, Endoscopic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EST in common bile duct stones (Active Comparator): With routine EST surgery, the sphincter is cut open and stones are removed
  Interventions: Procedure: EST
- ECPP in common bile duct stones (Experimental): Common bile duct stones are removed after EST, and then ECPP is performed.
  Interventions: Procedure: EST; Procedure: ECPP

INTERVENTIONS:
Procedure: EST — Stones are taken by cutting the papillary sphincter
Procedure: ECPP — During ERCP, a generous biliary sphincterotomy (>1 cm) will be performed to facilitate large stone extraction by use of a lithotripsy basket and a stone extraction balloon. After all stone fragments were cleared from the bile duct, this group will undergo ECPP after EST. A single-pigtail biliary stent will be placed (suspended overlength biliary stent, 7F × 20 cm). Then the rotatable repeatable opening and closing of soft tissue clamps (referred to as harmony clips, Mico-Tech, ROCC-D-26-195) should be applied to extend the bile duct axially, linear clamp the incised duodenal papilla, taking care to avoid clamping the bile duct stent, and removing the bile duct stent 3 weeks after ECPP.
  Arms: ECPP in common bile duct stones

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) combined with endoscopic papillary sphinctomy (EST) is the preferred clinical treatment for common bile duct stones, and this minimally invasive treatment technique has been widely used in clinical practice for decades. However, even after successful stone removal by EST combined with various methods, the incidence of postoperative recurrent bile duct stones can still be as high as 9.8%~30% . The emergence of these long-term complications after EST surgery is currently thought to be related to the loss of Oddi sphincter function. In clinical practice, the investigators tried a new method to repair the Oddi sphincter, that is, after ERCP+EST stone removal, a metal clip was inserted into the endoscopic clamp through the duodenoscopy, and clamp precisely on both lateral edges of the nipple after incision. This procedure is called endoscopic nipple clipping (ECPP). Initial explorations in animal and human trials showed good results, with 3 weeks after clipping of the incised nipple not only showing scar repair of the nipple shape and structure, but also confirmed the recovery of sphincter function by Oddi sphincter manometry, the Oddi's sphincter basal pressure, contraction frequency and contraction amplitude were able to return to the pre-EST level. In summary, the investigators designed a single-center randomized controlled trial to explore and verify the clinical effect of ECPP on the prevention of recurrent bile duct stones within one year by comparing the incidence of recurrent bile duct stones within one year after EST surgery. By observing the changes of intestinal biliary reflux, biliary bacterial colonization, biliary microecology and bile metabolism after EST surgery, the pathogenesis of long-term complications such as recurrent bile duct stones after EST surgery was further sought.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) combined with endoscopic papillary sphinctomy (EST) is the preferred clinical treatment for common bile duct stones, and this minimally invasive treatment technique has been widely used in clinical practice for decades. However, even after successful stone removal by EST combined with various methods, the incidence of postoperative recurrent bile duct stones can still be as high as 9.8%~30% . The emergence of these long-term complications after EST surgery is currently thought to be related to the loss of Oddi sphincter function. EST sphincterotomy results in destruction of the Oddi sphincter structure, which in turn causes dysfunction and reflux of intestinal contents into the biliary tract (biliary reflux). In clinical practice, the investigators tried a new method to repair the Oddi sphincter, that is, after ERCP+EST stone removal, a metal clip was inserted into the endoscopic clamp through the duodenoscopy, and clamp precisely on both lateral edges of the nipple after incision. Initial explorations in animal and human trials showed good results, with 3 weeks after clipping of the incised nipple not only showing scar repair of the nipple shape and structure, but also confirmed the recovery of sphincter function by Oddi sphincter manometry, the Oddi's sphincter basal pressure, contraction frequency and contraction amplitude were able to return to the pre-EST level.

the investigators designed a single-center randomized controlled trial to explore and verify the clinical effect of ECPP on the prevention of recurrent bile duct stones within one year by comparing the incidence of recurrent bile duct stones within one year after EST surgery. This prospective study will be performed at 1 tertiary hospitals in China. The investigators will recruit patients according to admission criteria and exclusion criteria. The patients will be randomized (at a 1:1 ratio) to endoscopic papillary sphinctomy (EST) group (control group) and endoscopic nipple clipping (ECPP) group (experimental group). The control groups will be followed by routine EST stone removal, the patient's postoperative nipple is in a post-incision state; The experimental group underwent ECPP after EST. The primary endpoint is the incidence of recurrent bile duct stones. The secondary outcomes include the mortality of each group, adverse events and the rate of technical success.

ELIGIBILITY:
Inclusion Criteria:

* Imaging confirms the presence of common bile duct stones.
* Common bile duct stones ≥ 1.0 cm in length.
* Common bile duct inner diameter≥1.2cm.
* The patient agrees to participate in the trial and signs the informed consent form.

Exclusion Criteria:

* Combined with coagulation dysfunction.
* heart, lung, kidney or other serious organic diseases.
* Patients with severe psychiatric illness.
* Previous papillary sphincterotomy.
* Patients who cannot cooperate with the completion of this study.
* Those with a life expectancy of less than 1 year and may not be able to complete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent bile duct stones | 12 months after ERCP
  The patient developed a recurrence of common bile duct stones within 1 year after surgery. Signs of recurrent bile duct stones include symptoms of cholangitis such as abdominal pain, fever, jaundice, or re-elevation of direct bilirubin/GGT/ALP or simple imaging of common bile duct stones.

SECONDARY OUTCOMES:
Death or adverse events | 12 months after ERCP
  The patient dies or develops postoperative complications of ERCP, stent displacement, detachment, etc., failure of ERCP.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, archiater, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kageoka M, Watanabe F, Maruyama Y, Nagata K, Ohata A, Noda Y, Miwa I, Ikeya K. Long-term prognosis of patients after endoscopic sphincterotomy for choledocholithiasis. Dig Endosc. 2009 Jul;21(3):170-5. doi: 10.1111/j.1443-1661.2009.00880.x. PMID 19691764
- [Background] Nzenza TC, Al-Habbal Y, Guerra GR, Manolas S, Yong T, McQuillan T. Recurrent common bile duct stones as a late complication of endoscopic sphincterotomy. BMC Gastroenterol. 2018 Mar 15;18(1):39. doi: 10.1186/s12876-018-0765-3. PMID 29544453
- [Background] Tanaka M, Takahata S, Konomi H, Matsunaga H, Yokohata K, Takeda T, Utsunomiya N, Ikeda S. Long-term consequence of endoscopic sphincterotomy for bile duct stones. Gastrointest Endosc. 1998 Nov;48(5):465-9. doi: 10.1016/s0016-5107(98)70086-0. PMID 9831833
- [Background] Yang J, Jin H, Gu W, Zhang X, Zhang X. Determinants of long-term complications of endoscopic sphincterotomy are infections and high risk factors of bile duct and not sphincter of Oddi dysfunction. Eur J Gastroenterol Hepatol. 2015 Apr;27(4):412-8. doi: 10.1097/MEG.0000000000000295. PMID 25874514
- [Background] Costamagna G, Tringali A, Shah SK, Mutignani M, Zuccala G, Perri V. Long-term follow-up of patients after endoscopic sphincterotomy for choledocholithiasis, and risk factors for recurrence. Endoscopy. 2002 Apr;34(4):273-9. doi: 10.1055/s-2002-23632. PMID 11932781
- [Background] Sugiyama M, Atomi Y. Risk factors predictive of late complications after endoscopic sphincterotomy for bile duct stones: long-term (more than 10 years) follow-up study. Am J Gastroenterol. 2002 Nov;97(11):2763-7. doi: 10.1111/j.1572-0241.2002.07019.x. PMID 12425545
- [Background] Mortensen FV, Jepsen P, Tarone RE, Funch-Jensen P, Jensen LS, Sorensen HT. Endoscopic sphincterotomy and long-term risk of cholangiocarcinoma: a population-based follow-up study. J Natl Cancer Inst. 2008 May 21;100(10):745-50. doi: 10.1093/jnci/djn102. Epub 2008 May 13. PMID 18477806
- [Background] Stromberg C, Luo J, Enochsson L, Arnelo U, Nilsson M. Endoscopic sphincterotomy and risk of malignancy in the bile ducts, liver, and pancreas. Clin Gastroenterol Hepatol. 2008 Sep;6(9):1049-53. doi: 10.1016/j.cgh.2008.04.016. Epub 2008 Jun 30. PMID 18585972
- [Background] Afghani E, Lo SK, Covington PS, Cash BD, Pandol SJ. Sphincter of Oddi Function and Risk Factors for Dysfunction. Front Nutr. 2017 Jan 30;4:1. doi: 10.3389/fnut.2017.00001. eCollection 2017. PMID 28194398
- [Background] Mandryka Y, Klimczak J, Duszewski M, Kondras M, Modzelewski B. [Bile duct infections as a late complication after endoscopic sphincterotomy]. Pol Merkur Lekarski. 2006 Dec;21(126):525-7. Polish. PMID 17405290
- [Background] Yasuda I, Fujita N, Maguchi H, Hasebe O, Igarashi Y, Murakami A, Mukai H, Fujii T, Yamao K, Maeshiro K, Tada T, Tsujino T, Komatsu Y. Long-term outcomes after endoscopic sphincterotomy versus endoscopic papillary balloon dilation for bile duct stones. Gastrointest Endosc. 2010 Dec;72(6):1185-91. doi: 10.1016/j.gie.2010.07.006. Epub 2010 Sep 25. PMID 20869711
- [Background] Wang Y, Chang H, Zhang Y, Wang K, Zhang H, Yan X, Meng L, Yao W, Li K, Huang Y. Endoscopic endoclip papilloplasty preserves sphincter of oddi function. Eur J Clin Invest. 2021 Mar;51(3):e13408. doi: 10.1111/eci.13408. Epub 2020 Sep 22. PMID 32929751